CLINICAL TRIAL: NCT01703403
Title: Physical Therapy Management in Degenerative Lumbar Diseases and Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201205036RIC
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Low Back Pain
Keywords: physical therapy; treated at NTUH and received rehabilitation at the PTC in recent ten years.
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Low back pain is a common health issue in elderly population. According to the statistics, more than 80% of Taiwanese suffer low back pain in the life. The cause of low back pain includes lumbar spondylosis, osteoporosis, compression fracture, muscle strain, spondylolisthesis…etc. In addition to drugs and surgery, physical therapy is an alternative choice for conservative treatment. Therefore, in this study, the investigators propose to analyze the physical examination, diagnostic methods, X ray, physical therapy records, physical therapy methods and clinical outcomes in patients with the diagnosis including lumbar spondylosis, low back pain, osteoporosis, compression fracture, back pain treated at National Taiwan University Hospital and received rehabilitation at the Physical Therapy Center in recent ten years.

ELIGIBILITY:
Experimental group:

Inclusion Criteria:

* patients with the diagnosis including lumbar spondylosis, low back pain, osteoporosis, compression fracture, back pain treated at National Taiwan University Hospital
* received rehabilitation at the Physical Therapy Center in recent ten years.

Control group:

Inclusion Criteria:

* patients with the diagnosis including lumbar spondylosis, low back pain, osteoporosis, compression fracture, back pain treated at National Taiwan University Hospital
* not received rehabilitation at the Physical Therapy Center in recent ten years.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with the diagnosis including lumbar spondylosis, low back pain, osteoporosis, compression fracture, back pain treated at National Taiwan University Hospital and received rehabilitation at the Physical Therapy Center in recent ten years.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-05

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PT,PhD, Principal Investigator — School of physical therapy, National Taiwan University
Locations (1):
- School & Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan